CLINICAL TRIAL: NCT05595473
Title: A Phase 1/2a, Open-label, Multicenter, Dose Escalation and Dose Expansion Study Evaluating the Safety, Tolerability and Efficacy of RZ-001 in Combination with Valganciclovir in Subjects with Hepatocellular Carcinoma
Brief Title: A Study to Evaluate the Safety, Tolerability and Efficacy of RZ-001 with Valganciclovir (VGCV) in Subjects with Hepatocellular Carcinoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rznomics, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RZ-001
Record Dates: First submitted 2022-09-07; First posted 2022-10-27 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 (Experimental)
  Interventions: Drug: RZ-001 Dose 1
- Cohort 2 (Experimental)
  Interventions: Drug: RZ-001 Dose 2
- Cohort 3 (Experimental)
  Interventions: Drug: RZ-001 Dose 3
- Cohort 4 (Experimental)
  Interventions: Drug: RZ-001 Dose 4

INTERVENTIONS:
Drug: RZ-001 Dose 1 — RZ-001 Dose 1 and VGCV
  Arms: Cohort 1
Drug: RZ-001 Dose 2 — RZ-001 Dose 2 and VGCV
  Arms: Cohort 2
Drug: RZ-001 Dose 3 — RZ-001 Dose 3 and VGCV
  Arms: Cohort 3
Drug: RZ-001 Dose 4 — RZ-001 Dose 4 and VGCV
  Arms: Cohort 4

SUMMARY:
This is first in human study to evaluate the safety, tolerability, immunogenicity, and preliminary clinical activity of RZ-001 when given to subjects with human telomerase reverse transcriptase (hTERT)-positive HCC.

DETAILED DESCRIPTION:
The study will be conducted in 2 parts.

Part 1 is a dose escalation study which aims to explore the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) after the single escalating dose of the intratumoral (IT) injection given through 4 different cohorts.

Part 2 will consist of dose expansion, exploring clinical activity for the optimal fixed dose based on the results of Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females
* Hepatocellular carcinoma diagnosis (BCLC stage B or C)
* hTERT positive expression confirmed during the screening period
* ECOG score of 0 or 1
* Child-Pugh score of A to B7
* Life expectancy >= 3 months

Exclusion Criteria:

* Moderate or severe ascites
* History of hepatic encephalopathy
* Carcinomas other than HCC
* Current or history of HIV positive
* Not suitable for inclusion judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose limiting toxicities (DLT) in Part 1 as graded by NCI-CTCAE | Day 1 to Day 28
To determine safety and efficacy of RZ-001 by changes in overall response rate (ORR) for participants in part 2 as graded by RECIST v1.1 and mRECIST | Day 1 to Day 15
To determine safety and efficacy of RZ-001 by changes in duration of response (DOR) in part 2 as graded by RECIST v1.1 and mRECIST | Day 1 to Day 15
To determine safety and efficacy of RZ-001 by changes in Progression free survial (PFS) of participants in part 2 as graded by RECIST v1.1 and mRECIST | Day 1 to Day 15
To determine safety and efficacy of RZ-001 by changes in overall survival (OS) of participants in part 2 as graded by RECIST v1.1 and mRECIST | Day 1 to Day 15
Number of participants with adverse events (AEs) in part 1 and 2 as graded by NCI-CTCAE | Day 1 to Day 28

SECONDARY OUTCOMES:
To determine safety and efficacy of RZ-001 by changes in overall response rate (ORR) of the partipants in Part 1 as graded by RECIST v1.1 and mRECIST | Day 1 to Day 15
To determine safety and efficacy of RZ-001 by changes in duration of response (DOR) of the partipants in Part 1 as graded by RECIST v1.1 and mRECIST | Day 1 to Day 15
To determine safety and efficacy of RZ-001 by changes in Progression free survial (PFS) of the partipants in Part 1 as graded by RECIST v1.1 and mRECIST | Day 1 to Day 15
To determine safety and efficacy of RZ-001 by changes in overall survival (OS) of the partipants in Part 1 as graded by RECIST v1.1 and mRECIST | Day 1 to Day 15

CONTACTS AND LOCATIONS:
Locations (5):
- South Korea (5):
  - Samsung Medical Center, Seoul, Seoul
  - Kyungpook National University Hospital, Deagu
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No